CLINICAL TRIAL: NCT01676324
Title: FOCUS: The Future of Fecal Calprotectin Utility Study for the Diagnosis and Management of IBD
Brief Title: FOCUS: The Future of Fecal Calprotectin Utility Study for the Diagnosis and Management of Inflammatory Bowel Disease (IBD)
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H12-01499
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Fecal Calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: Those with Inflammatory Bowel Disease (known) and those with no Inflammatory Bowel Disease (not previously diagnosed)

SUMMARY:
Hypothesis:

Fecal Calprotectin will be useful in guiding the diagnosis and management of patients with Inflammatory Bowel Disease. Fecal Calprotectin can be utilized as an alternative to colonoscopy in the management of patients with Inflammatory Bowel Disease.

Objectives:

By means of a survey from the ordering physician we would assess:

Primary Endpoint

1. The Percentage of time that the Fecal Calprotectin result caused the physician to change the management of a patient.

Secondary Endpoints

1. To determine if the Fecal Calprotectin result influenced the number of endoscopies performed
2. To correlate how well the Fecal Calprotectin correlates with Endoscopic findings when endoscopy was performed.
3. To assess the correlation between the Fecal Calprotectin level and symptoms as measured by the Harvey Bradshaw index or the partial Mayo Score (or full Mayo Score depending if endoscopy was performed).

DETAILED DESCRIPTION:
Patients will be identified as eligible by the attending Gastroenterologist during the course of a usual consultation. Patients will be referred to the research nurse in the doctor's office for further information regarding the study and informed consent will be obtained by the research nurse.

Upon enrollment, the physician or the research nurse will complete an online requisition form with a unique code which will provide the baseline data. The patient will be provided with the Easy Sampler™ collection kit and instructions on the use of this kit and location on where to send the specimen.

The nurse will then send an email to the research nurse in the originating physician's office with the result of the calprotectin assay. The research nurse will review the result with the physician. After physician review, either the physician or the research nurse will then complete a follow up survey online.

After completion of the assays and surveys, the data will be tabulated electronically from the online website and analyzed by the PI and/or co-investigators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 19 years of age or older, they must be able to read and provide written consent in English.

Subjects will have gastrointestinal symptoms or be known to have Inflammatory Bowel Disease whereby the clinician feels that obtaining Fecal Calprotectin may be useful in the care of the patient. Patients must be able to collect a feces sample and return it for analysis within 3 days

Exclusion Criteria:

* Known Ischemic colitis, infectious enteritis or colitis, known colorectal cancer, history of extensive bowel resection, ostomy, current daily use of NSAIDs (aspirin, ibuprofen, naproxen, etc) or the inability to collect sample and return it within 3 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be those age 19 or older seen by community and academic gastroenterologists and may be referred for Fecal Calprotectin testing at the discretion of the Gastroenterologist.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of time that Fecal Calprotectin result caused the physician to change the management of a patient. | one year
  The utility of the test will be assessed by comparing the proportion of time the test altered management for each of the two groups (IBD present vs. IBD absent). The groups will be compared using paired t-tests and McNemar's test as appropriate. Multivariate analysis will be used to assess the impact of the baseline variables on the test utility.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, Principal Investigator — Department of Medicine, Division of Gastroenterology, UBC
Locations (1):
- GI Research Institute (GIRI), Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Sutherland AD, Gearry RB, Frizelle FA. Review of fecal biomarkers in inflammatory bowel disease. Dis Colon Rectum. 2008 Aug;51(8):1283-91. doi: 10.1007/s10350-008-9310-8. Epub 2008 Jun 10. PMID 18543035
- [Background] Gisbert JP, Bermejo F, Perez-Calle JL, Taxonera C, Vera I, McNicholl AG, Algaba A, Lopez P, Lopez-Palacios N, Calvo M, Gonzalez-Lama Y, Carneros JA, Velasco M, Mate J. Fecal calprotectin and lactoferrin for the prediction of inflammatory bowel disease relapse. Inflamm Bowel Dis. 2009 Aug;15(8):1190-8. doi: 10.1002/ibd.20933. PMID 19291780
- [Background] Schoepfer AM, Beglinger C, Straumann A, Trummler M, Vavricka SR, Bruegger LE, Seibold F. Fecal calprotectin correlates more closely with the Simple Endoscopic Score for Crohn's disease (SES-CD) than CRP, blood leukocytes, and the CDAI. Am J Gastroenterol. 2010 Jan;105(1):162-9. doi: 10.1038/ajg.2009.545. Epub 2009 Sep 15. PMID 19755969
- [Result] Keohane J, O'Mahony C, O'Mahony L, O'Mahony S, Quigley EM, Shanahan F. Irritable bowel syndrome-type symptoms in patients with inflammatory bowel disease: a real association or reflection of occult inflammation? Am J Gastroenterol. 2010 Aug;105(8):1788, 1789-94; quiz 1795. doi: 10.1038/ajg.2010.156. Epub 2010 Apr 13. PMID 20389294